CLINICAL TRIAL: NCT01091337
Title: Comparative Study on the Efficacy and Safety of Procaterol vs Salbutamol Given Via Metered Dose Inhaler With Spacer in the Management of Acute Asthma Attack in the Emergency Room
Brief Title: Comparative Study on the Efficacy and Safety of Procaterol Versus Salbutamol Given Via Metered Dose Inhaler With Spacer in the Management of Acute Asthma Attack in the Emergency Room
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical, Inc., Philippines (Industry)
Responsible Party: Dr. Camilo Roa, MD / Study Principal Investigator, Philippine General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOIAA-MPT-2005-01
Record Dates: First submitted 2010-03-05; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Procaterol; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Procaterol (Experimental): Procaterol(Meptin Air) MDI, 20 ug or 2 puffs every 20 minutes
  + Hydrocortisone, 100 mg IV shall be given immediately at start of treatment
  Interventions: Drug: Procaterol
- Salbutamol (Active Comparator): Salbutamol(Ventolin Inhaler) MDI, 40 ug or 4 puffs every 20 minutes + Hydrocortisone, 100 mg IV shall be given immediately at start of treatment
  Interventions: Drug: Salbutamol

INTERVENTIONS:
Drug: Procaterol — Procaterol(Meptin Air) MDI, 20 ug or 2 puffs every 20 minutes
  + Hydrocortisone, 100 mg IV shall be given immediately at start of treatment
  Other Names: Meptin Air
  Arms: Procaterol
Drug: Salbutamol — Salbutamol(Ventolin Inhaler) MDI, 40 ug or 4 puffs every 20 minutes + Hydrocortisone, 100 mg IV shall be given immediately at start of treatment
  Other Names: Ventolin Inhaler
  Arms: Salbutamol

SUMMARY:
To compare the efficacy and safety of inhaled procaterol (Meptin Air) versus inhaled salbutamol as metered dose inhaler (MDI) reliever of acute exacerbation of asthma not in imminent respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 20 years old and above who are brought to the Emergency Room (ER) with acute bronchospasm
* Diagnosed cases of bronchial asthma based on history, physical examination and pulmonary function test
* Patients maintained on inhaled steroids who have no active medical problems (such as pulmonary TB, cardiac and renal diseases) aside from asthma
* Presence of known risk factors for asthma mortality does not disqualify patients from the study unless they are in impending respiratory failure
* All patients must sign the informed consent form

Exclusion Criteria:

* Patients who are in respiratory distress consistent with severe exacerbation requiring intensive care hospital admission
* Who had intake of oral bronchodilator 6 hrs prior to consult
* Who had intake of oral steroids within the last 24 hrs
* Those with positive history of allergy and hypersensitivity to procaterol and salbutamol
* Patients who are diagnosed or clinically suspected to have COPD (ever-smokers with >10 pack-years smoking history or those exposed to workplaces where there is a heavy smoke load)
* Presence of concurrent disease/diseases that may aggravate asthma thereby delaying bronchodilator response (e.g., pneumonia, pulmonary congestion and others)
* Patients with other medical conditions which are serious enough to warrant immediate concurrent therapy during the 1 hour study and/or whose condition can be adversely affected by the treatment given (like uncontrolled diabetes, renal failure and hepatic insufficiency)
* The NIH Working Group on Asthma and Pregnancy has recommended that pregnant asthmatics are treated as aggressively as non-pregnant patients particularly during acute asthmatic attack. , Bronchodilators (except for epinephrine which is not in this study) have been found safe in pregnancy with a risk class of B and C. For these reasons, pregnancy by itself is not an exclusion criterion in this study and a pregnancy test will not be required for those who are in the childbearing age group. Requiring the test will unnecessarily delay the treatment for acute asthma. However, those who are suspected to be suffering from pregnancy-related complications like vaginal bleeding, premature labor, pre-eclampsia and others, are excluded.
* Severe Acute Asthma Attack, a reason for patient exclusion, shall be defined in this study as the presence of any one of the following criteria:

  1. Severe asthma with a lack of response to initial therapy in the emergency department or worsening asthma despite adequate therapy.
  2. Presence of confusion, drowsiness, other signs of impending respiratory arrest, or loss of consciousness
  3. Wood-Downe's clinical asthma scoring score of >5 (see table 2 below)
* Any patient who is currently participating in other drug trials and/or having participated in other drug trials for less than 1 month of termination of the trial are excluded
* Patients who have previously participated in this study are excluded

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2006-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the bronchodilator efficacy of inhaled procaterol (Meptin Air) vs. inhaled salbutamol used as MDI reliever of acute exacerbation of asthma in the ER. | < 12 hours

SECONDARY OUTCOMES:
To evaluate the safety of procaterol MDI (Meptin Air) versus salbutamol MDI in the management of acute exacerbation of asthma in terms of adverse side effects such as palpitations, tachycardia, tremor, and hypokalemia. | < 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Camilo Roa, MD, Principal Investigator — Philippine General Hospital
Locations (1):
- Philippine General Hospital, Manila, Philippines